CLINICAL TRIAL: NCT00990379
Title: Cellular and Molecular Kinetics of Cerebrospinal Fluid (CSF) Using Heavy Water Labeling Method: A Study of Healthy Controls, CNS HIV Infection, Parkinson's Disease and Other Neurodegenerative Diseases
Brief Title: Using Heavy Water to Study Cell Dynamics in Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Salena Killion (Industry)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor-Investigator, Salena Killion, Director of Clinical Studies, KineMed
Organization: KineMed (Industry)
Other Study IDs: 6076
Record Dates: First submitted 2009-10-02; First posted 2009-10-06 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Parkinson's Disease; HIV Infections
Keywords: HIV; brain diseases; spinal fluid; HIV positive
MeSH Terms: conditions — Parkinson Disease; HIV Infections; Brain Diseases; HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Controls: Healthy men and women, 18 years of age or older, who have no history of significant medical conditions.
- HIV positive: Men and women, 18 years of age or older, who have been diagnosed with HIV infection. Patients may be on or off of ARVs.
- Parkinson's Disease: Men and women, 18 years of age or older, who have been diagnosed with Parkinson's Disease.

SUMMARY:
This pilot study will assess the feasibility of using heavy water as a safe 'tracer' for biomarker studies of diseases of the brain and spinal cord, that, together, are also called the central nervous system (CNS). Heavy water, also called deuterated water or D20, is the same as normal drinking water except the hydrogen atoms have been replaced by deuterium, a naturally occurring isotope of hydrogen. In particular, this study will use heavy water to define: 1) The rate of immune cell proliferation (growth) in the cerebrospinal fluid (CSF) compared to blood. This study will be examining a particular type of immune cell called T lymphocytes. 2) This study will also examine selected molecules generated by nerve cells of the CNS to understand their rate of secretion and turnover in healthy control participants, HIV-1-infected participants and participants with a non-HIV-related neurodegenerative disease such as Parkinson's disease (PD).

This study will involve the administration of heavy water orally for either seven days, 12 days or six weeks. Measurements will be taken by lumbar puncture (LP, also known as a spinal tap). Blood (approximately five tablespoons per visit) will also be obtained at each of the lumbar puncture appointments.

If this method can be used to establish the rates of immune cell turnover and the production rates of neuronal molecules using cerebrospinal fluid, it will provide unique data that is important to understand chronic neurodegenerative conditions, like PD, and to measure responses to targeted therapies.

Hypothesis:

1. D2O, administered orally, can be used to measure the proliferation rates of CSF T cells (and, eventually, of their major phenotypic subsets).
2. D2O can be used to assess the turnover and production rates of CNS constituents that are normally or pathologically shed or secreted into the CSF, including (eventually): cargo molecules transported specifically in neurons in the CNS, such as chromogranin-A and -B, neuregulin-1 (specifically the extracellular secreted ectodomain of neuronal differentiation factor (NDF) isoform type α1, α2, β1, and the acetylcholine receptor inducing activity isoform (ARIA), secreted amyloid precursor protein (sAPP), alpha-synuclein; and APP metabolites amyloid beta (Aβ) 41 and 42.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* healthy controls with no significant medical conditions
* diagnosed HIV positive patients on or off ARVs
* diagnosed Parkinson's Disease patients
* capacity to provide informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy controls, HIV positive (on or off ARVs), patients diagnosed with Parkinson's Disease.
  All subjects must be 18 years of age or older.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2009-04; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
CSF Biomarkers | 40 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard Price, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States